CLINICAL TRIAL: NCT05422885
Title: Senolytics To Alleviate Mobility Issues and Neurological Impairment in Aging
Brief Title: Safety and Feasibility of Dasatinib and Quercetin in Adults at Risk for Alzheimer's Disease
Acronym: STAMINA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lewis Lipsitz (Other)
Responsible Party: Sponsor-Investigator, Lewis Lipsitz, Director, Marcus Institute for Aging Research, Hebrew SeniorLife
Organization: Hebrew SeniorLife (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00053594
Record Dates: First submitted 2022-03-14; First posted 2022-06-21 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Aging
Keywords: Alzheimer's disease; Senescence
MeSH Terms: conditions — Alzheimer Disease | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Dasatinib and Quercetin
  Interventions: Drug: Dasatinib; Drug: Quercetin

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 100 mg for 2 consecutive days, every two weeks for 12 weeks
  Other Names: Sprycel
Drug: Quercetin — Quercetin 1,250 mg for 2 consecutive days, every two weeks for 12 weeks

SUMMARY:
The purpose of this pilot study is to demonstrate the safety and feasibility of administering intermittent doses of Dasatinib and Quercetin (D+Q) in older adults at risk of Alzheimer's disease (AD). The study will evaluate whether giving D+Q may improve cerebral blood flow regulation, mobility, and cognition in older adults, and thus may prevent progression to Alzheimer's disease.

DETAILED DESCRIPTION:
The investigators will conduct a 12-week single arm, open label, pre-post pilot study in 12 adults aged 65 or older with slow gait speed (<1.0 m/sec) and Mild Cognitive Impairment (MCI, defined as a Telephone Montreal Cognitive Assessment Score (MoCA) <19). Participants will be asked to take 100mg of Dasatinib and 1,250mg of Quercetin for 2 consecutive days, every two weeks over a period of 12 weeks (12 doses in total, given over 6 cycles).

At baseline, enrolled participants will undergo gait speed and neurocognitive testing, and provide blood and urine to evaluate biomarkers of senescence. At visits 3,4, 6, and 7, participants will have safety labs drawn, and the study team will assess medication adherence and adverse events. At visits 2, 5, and 8, participants will undergo cognitive assessments, gait speed testing, cerebral blood flow and neurovascular coupling testing. At the final study visit, participants will again provide blood and urine to assess biomarkers of senescence.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >/= 65 years
* Ambulatory,
* Community dwelling,
* Slow gait speed (<1 m/second),
* Mild Cognitive Impairment (Telephone MoCA score <21, which is indicative of cognitive impairment)

Exclusion Criteria, or as per clinical judgment:

* Telephone MoCA score <10 points
* Unwilling to take study medications or follow study protocol
* Inability to independently perform Katz Activities of Daily Living (ADLs),
* Allergies to Dasatinib or Quercetin,
* Hospitalization within 6 months,
* Unstable coronary artery disease (myocardial infarction within 6 months or angina),
* Stroke or transient ischemic attack in the past 6 months,
* Chronic heart failure,
* Current or chronic history of liver disease,
* Neurodegenerative disease including Parkinson's disease,
* Anemia,
* Chronic renal disease,
* Drug or alcohol abuse in the last 5 years,
* QTc prolongation,
* Thrombocytopenia,
* Neutropenia,
* Prolonged prothrombin time or INR,
* Indications of current fluid retention,
* History or current diagnosis of pulmonary hypertension,
* Inability to insonate the middle cerebral artery through a temporal bone window on at least one side using transcranial Doppler ultrasound, or
* Chronic use of any of the following medications: anti-arrhythmic medications, antipsychotics, anxiolytics, anti-platelet or anti-coagulant medications other than aspirin, quinolone antibiotics, or drugs metabolized by the same liver enzymes as Quercetin or Dasatinib.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Lipsitz, MD, Principal Investigator — Hebrew Senior Life
Locations (1):
- Hebrew Senior Life, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Millar CL, Iloputaife I, Baldyga K, Kuo J, Tchkonia T, Kirkland JL, Travison TG, Lipsitz LA. Rationale and Design of STAMINA: Senolytics To Alleviate Mobility Issues and Neurological Impairments in Aging, A Geroscience Feasibility Study. Transl Med Aging. 2023;7:109-117. doi: 10.1016/j.tma.2023.10.004. Epub 2023 Oct 21. PMID 40248131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 2022-2024 in the greater Boston, MA area. Individuals were recruited through a recruitment firm that utilizes online targeted advertisements based on an individual's browsing history, as well as senior housing presentations, study flyers at clinical practices, and invitations to previous research volunteers who agreed to be in our participant registries.
Pre-assignment Details: Of the 332 individuals that expressed interest in the study, 115 were screened via telephone. Sixty were ineligible due to not meeting the pre-specified inclusion/exclusion criteria. Of the 55 eligible telephone screeners, 24 were not enrolled due to loss of interest (n=12), loss to follow-up (n=10), or closed enrolment (n=2). Of the 31 participants that were screened in-person, 16 were excluded for various reasons, while 15 individuals were eligible and willing to participate.
Groups:
- Dasatinib and Quercetin: Participants took 100 mg of Dasatinib and 1,250 mg of Quercetin for 2 consecutive days, every two weeks for 12 weeks
Period: Overall Study
Arm/Group | Dasatinib and Quercetin
Started | 15
Completed | 12
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Highest Level of Education [Count of Participants; unit: Participants]
  No Diploma | 1
  Some College/Vocational School | 1
  Associates Degree | 1
  Bachelors Degree | 5
  Graduate/Doctoral/Law Degree | 7
4-meter Gait Speed [Mean (Standard Deviation); unit: meters/second] | 0.8 (0.1)
Telephone Montreal Cognitive Assessment Score [Mean (Standard Deviation); unit: points] — Range: 0-22 points with higher scores indicating higher cognitive status
  points | 17 (2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27 (4)
Osteo- or Degenerative Arthritis [Count of Participants; unit: Participants] | 6
High Blood Pressure [Count of Participants; unit: Participants] | 5
High Cholesterol [Count of Participants; unit: Participants] | 6
Depression [Count of Participants; unit: Participants] | 4
Eye Disease [Count of Participants; unit: Participants] | 8
Stomach Disease (e.g., Acid Reflux) [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Neurovascular Coupling
Description: Change in cerebral blood flow during an N-back cognitive task using transcranial doppler ultrasound.
Time Frame: Screening, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
cm/s
  Screening | 0.68 (1.40)
  Week 8 | 0.26 (2.04)
  Week 14 | 0.80 (2.13)

2. Primary Outcome: Executive Function
Description: Assess change in executive cognitive function using TRAILS test, corrected for response time. Higher scores indicate worse executive functioning.
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
seconds
  Baseline (Week 2) | 80.6 (80.2)
  Week 8 | 75.0 (61.4)
  Week 14 | 63.4 (44.6)

3. Primary Outcome: Gait Speed
Description: Assess change in gait speed. Performed without a distracting cognitive task.
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
meters/second
  Baseline (Week 2) | 0.87 (0.15)
  Week 8 | 0.85 (0.16)
  Week 14 | 0.87 (0.14)

4. Primary Outcome: Montreal Cognitive Assessment (MoCA) Score
Description: The Montreal Cognitive Assessment evaluates global cognition. Scores range from 0-30 points, with higher scores indicating better cognition
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Arm 1
Number analyzed (Participants) | 12
points
  Baseline | 23 (2)
  8 Weeks | 25 (3)
  14 Weeks | 24 (2)

5. Secondary Outcome: Physical Performance
Description: Assessment of overall physical function using the short physical performance battery (SPPB) scored from 0-12, based on a composite of balance, strength, and walking speed. Higher scores indicate better mobility.
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
points
  Baseline (Week 2) | 9 (1)
  Week 8 | 9 (2)
  Week 14 | 9 (2)

6. Secondary Outcome: Mobility
Description: Test of mobility using timed up and go test, including standing from a chair, walking, and turning.
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
seconds
  Baseline (Week 2) | 14.2 (2.6)
  Week 8 | 13.9 (3.1)
  Week 14 | 13.6 (2.4)

7. Secondary Outcome: Grip Strength
Description: Measure of grip strength using a hand dynamometer.
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
kilograms
  Baseline (Week 2) | 23.5 (7.2)
  Week 8 | 22.7 (5.8)
  Week 14 | 23.6 (5.3)

8. Secondary Outcome: Gait Speed During Cognitive Task
Description: Measure of gait speed during a cognitive task.
Time Frame: Baseline, 8, and 14 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
meters/second
  Baseline (Week 2) | 0.76 (0.13)
  Week 8 | 0.75 (0.16)
  Week 14 | 0.78 (0.14)

9. Secondary Outcome: P16 ink4a Expression in CD3 Positive Cells
Description: Measure of P16 ink4a expression in senescent CD3 lymphocytes in the blood.
Time Frame: Screening and 14 weeks
Measure: Mean (Standard Deviation); unit: relative expression to housekeeping gene
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 10
relative expression to housekeeping gene
  Screening | 10.6 (5.2)
  Week 14 | 9.4 (3.8)

10. Secondary Outcome: SASP Factors in Blood and Urine
Description: Measure of the senescence-associated biomarkers IL-1alpha picogram/mL and IL-6 picogram/mL.
Time Frame: Screening and 14 weeks
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
picograms/mL
  Serum IL1-alpha Screening | 664.5 (368.1)
  Serum IL1-alpha Week 14 | 742.2 (513.1)
  Serum IL-6 Screening | 3.6 (1.7)
  Serum IL-6 Week 14 | 2.8 (1.5)

11. Secondary Outcome: SASP Factors in Blood and Urine
Description: Measure of the senescence-associated biomarkers MMP-9 nanograms/mL and MMP-12 nanograms/mL.
Time Frame: Screening and 14 weeks
Measure: Mean (Standard Deviation); unit: nanograms/mL
Arm/Group | Dasatinib and Quercetin
Number analyzed (Participants) | 12
nanograms/mL
  Serum MMP-9 Screening | 458.5 (189.4)
  Serum MMP-9 Week 14 | 541.6 (454.4)

ADVERSE EVENTS:
Time Frame: For all participants, adverse events were collected during the entire 14 week study. We were collecting during the period of June 2022 to January 2024, which is approximately 1 year and 8 months.
Arm/Group | Dasatinib and Quercetin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib and Quercetin (N=15)
Serious Adverse Event (Injury, poisoning and procedural complications) | 1 (1) — Participant was bitten by family dog on both hands. Waited until next day to go to urgent care which told him to go to hospital emergency room. He was admitted one night (discharged November 12) and sent home with antibiotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib and Quercetin (N=15)
Headache (General disorders) | 4 (5)
Producing more urine than usual (Renal and urinary disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (4)
High Glucose (Metabolism and nutrition disorders) | 2 (3)
Low White Blood Cell Count (Blood and lymphatic system disorders) | 3 (6)
High Cystatin C Value (Renal and urinary disorders) | 1 (1)
Irregular Glomerular Filtration Rate (Renal and urinary disorders) | 1 (2)
Ankle Edema (General disorders) | 1 (1)
Basilar Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Irregular Heart Beat (Cardiac disorders) | 1 (1)
Muscle or Hip Pain (Injury, poisoning and procedural complications) | 2 (2)
Difficulty with Balance (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed Mood or Anxiety (Psychiatric disorders) | 2 (2)
Sore Throat (General disorders) | 1 (1)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (2)
Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
High Potassium (Blood and lymphatic system disorders) | 1 (1)
High Creatinine (Blood and lymphatic system disorders) | 2 (2)
Diarrhea or Loose Stool (Gastrointestinal disorders) | 5 (9)
Fluttering in Chest (Cardiac disorders) | 1 (1)
Loss of Appetite or Nausea (Gastrointestinal disorders) | 3 (8)
Fatigue or Tiredness (General disorders) | 6 (8)
Dizziness (General disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Low Hematocrit Level (Blood and lymphatic system disorders) | 1 (1)
Tingling in Extremeties (Nervous system disorders) | 1 (1)
Sprained wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Low blood pressure (Cardiac disorders) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Restless Sleep (General disorders) | 1 (1)
Memory Concerns (Psychiatric disorders) | 1 (1)
High Blood Urea Nitrogen (Renal and urinary disorders) | 1 (1)
High ALT Level (Hepatobiliary disorders) | 1 (1)
High Heart Rate (Cardiac disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Although we collected urine samples, the SASP factors (i.e., biomarkers) we were not measured due to insufficient funds and resources. Therefore, we are unable to analyze any data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT05422885/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05422885/SAP_001.pdf